CLINICAL TRIAL: NCT02516865
Title: Practical Approaches to Exercise in Moms
Acronym: PE Moms
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maxine Mendelson (Other)
Responsible Party: Sponsor-Investigator, Maxine Mendelson, Clinical Research Coordinator, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: IRB15-00117
Record Dates: First submitted 2015-05-13; First posted 2015-08-06 (Estimated); Last update posted 2015-08-06 (Estimated); Status verified 2015-08

CONDITIONS: Body Weight
Keywords: postpartum; physical activity
MeSH Terms: conditions — Body Weight; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Experimental)
  Interventions: Device: Fitbit activity tracker
- Group 2 (Experimental)
  Interventions: Device: Fitbit activity tracker; Device: Ankle weights
- Group 3 (No Intervention)

INTERVENTIONS:
Device: Fitbit activity tracker — Tracks steps taken, floors climbed, and distance traveled. Sleep quality is an additional measurement.
  Arms: Group 1; Group 2
Device: Ankle weights — Worn during typical daily activities.
  Arms: Group 2

SUMMARY:
This project aims to test the feasibility of a practical physical activity intervention for postpartum women, incorporating the use of body weights worn during typical daily activities.

DETAILED DESCRIPTION:
We are piloting a 3-arm, unblinded, randomized controlled trial in postpartum women; with 10 participants in each study group. Women will be recruited at 2-6 months postpartum, with the intervention lasting through 12 months postpartum. Data collection will include:1) Physical activity; 2) Maternal body composition; 3) Questionnaires to assess:motivation to adopt healthy behaviors, body attitudes, infant feeding practices; 4) Process evaluation to assess: likes and dislikes about the intervention program, suggestions for improving the intervention, reasons for leaving the study. The proposed study time period is 6 months for study recruitment, 18 months to carry out the study, and 6 months for data analysis (total 2 years).

ELIGIBILITY:
Inclusion Criteria:

* 2-6 months postpartum women

Exclusion Criteria:

* Premature birth
* History of serious illness
* Medically incapable of low-intensity exercise
* Currently taking medications that cause weight loss

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Change in baseline body weight at 12-months postpartum. | Baseline and 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States